CLINICAL TRIAL: NCT00201682
Title: Phase I/II Study of Etanercept and Rituximab in Patients With Chronic Lymphocytic Leukemia and Small Lymphocytic Lymphoma
Brief Title: Etanercept and Rituximab in Patients With Chronic Lymphocytic Leukemia and Small Lymphocytic Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: John Byrd (Other)
Responsible Party: Sponsor-Investigator, John Byrd, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-0113
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: Leukemia; Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia; Lymphoma | interventions — Etanercept; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Etanercept 25 mg administered sub-cutaneously twice weekly (Monday and Thursday) weeks 1-5 of therapy (total of 10 doses). The third dose of etanercept will be administered 1 hour prior to receiving rituximab. Rituximab: Patients will receive 375 mg/M2 of rituximab three times weekly for four weeks (a total of 12 doses of rituximab).
  Interventions: Drug: Etanercept; Drug: Rituximab

INTERVENTIONS:
Drug: Etanercept — 25 mg SQ twice weekly weeks 1-5
  Other Names: Enbrel
Drug: Rituximab — (375 mg/m2) Using Stepped-Up Dosing Thrice Weekly, weeks 2-5
  Other Names: RITUXAN®

SUMMARY:
This is a phase I/II study of the combination of etanercept and rituximab in patients with chronic lymphocytic leukemia (CLL) and small lymphocytic lymphoma (SLL). This combination is proposed to improve the efficacy and diminish the toxicity of this the

DETAILED DESCRIPTION:
Rationale: Previous research has demonstrated that rituximab has efficacy against chronic lymphocytic leukemia (CLL) and small lymphocytic lymphoma (SLL). Rituximab is a monoclonal antibody used to treat different types of lymphomas. Monoclonal antibodies are a type of immunotherapy used against some types of cancer. They are produced in a laboratory and designed to target as well as bind with cells that carry specific proteins. Rituximab attaches to a protein called CD20 that is found almost exclusively on the surface of B-cells. Once rituximab attaches to the protein, the immune system activates to kill the malignant B-cells. Researchers are investigating what other therapies to combine with rituximab to reduce side effects and improve patient outcomes. The current study combines etanercept with rituximab. Etanercept is an anti-inflammatory agent being tested as a therapy for cancer. Researchers want to assess the theory that etanercept may reduce the toxicity associated with rituximab in patients and increase efficacy while providing its own treatment benefit to patients.

Purpose: This study is evaluating the safety and efficacy of combination etanercept and rituximab in patients with CLL and SLL. The biological response of tumor cells and the immune system to this drug combination will also be measured in patients before, during, and after therapy administration.

Treatment: Patients in this study will receive etanercept and rituximab. Etanercept is given through injections into the skin and rituximab through intravenous infusions. During the first week of the study, etanercept alone will be given to patients two times. During the second week, patients will continue receiving etanercept twice weekly and begin receiving rituximab three times weekly. This schedule of etanercept twice weekly and rituximab three times weekly will be repeated four times. Several tests and exams will be given throughout the study to closely monitor patients. Treatments will be discontinued due to disease growth or unacceptable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Must have been previously treated CLL/SLL
* Must have CD20 expression
* ECOG PS =<3
* No prior Campath-1H
* No active infection requiring antibiotics
* No concurrent immunosuppressive therapy
* No prior history demyelinating neurologic disease
* No active viral hepatitis

Exclusion Criteria:

* No pregnant or breastfeeding women
* ECOG PS =4
* Life expectancy of >12 weeks
* Patients with bilirubin or creatinine>3.0 mg/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2002-10; Primary Completion 2006-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
To determine the feasibility and toxicity of the combination of etanercept and rituximab in patients with CLL/SLL. | up to 1 year
Determine if etanercept increases the complete response rate while decreasing the frequency of infusion-related toxicity in patients with CLL/SLL receiving rituximab therapy. | up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: John Byrd, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Result] Woyach JA, Lin TS, Lucas MS, Heerema N, Moran ME, Cheney C, Lucas DM, Wei L, Caligiuri MA, Byrd JC. A phase I/II study of rituximab and etanercept in patients with chronic lymphocytic leukemia and small lymphocytic lymphoma. Leukemia. 2009 May;23(5):912-8. doi: 10.1038/leu.2008.385. Epub 2009 Feb 19. PMID 19225537
- See also: Jamesline — http://cancer.osu.edu